CLINICAL TRIAL: NCT07142382
Title: Effect of Different Hip Bathing Methods on Perianal Abscess After Surgery: a Single-center, Prospective, Open-label Randomized Controlled Trial
Brief Title: Effect of Different Sitz Bath Methods on Perianal Abscess After Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PutianU-004
Record Dates: First submitted 2025-08-13; First posted 2025-08-26 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Perianal Abscess
Keywords: sitz bath; perianal absecess; Wound healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional group (No Intervention): Patients in the conventional group were advised to use a regular bidet without a flusher after surgery. The patient was treated with potassium permanganate sitz bath from the first postoperative day. The concentration of potassium permanganate solution used in the sitz bath was 0.02%. The patient had a sitz bath three times a day (9:00, 13:00, and 17:00) and the perianal area was scrubbed through a cotton cloth. Each sitz bath lasts 10-15 minutes and the water temperature is 41-43 ° C.
- Manual group (Experimental): Patients in the manual group were advised to use a manual flushing bidet with an irrigator after surgery. The patient was treated with potassium permanganate sitz bath from the first postoperative day. The concentration of potassium permanganate solution used in the sitz bath was 0.02%. The patients were advised to have a sitz bath three times a day (9:00, 13:00, 17:00). By manually pressing the airbag, the potassium permanganate solution in the bidet was sprayed with the rinsing device to achieve the purpose of cleaning the perianal area. The duration of each sitz bath was 10-15 minutes, and the water temperature was 41-43 ° C.
  Interventions: Behavioral: Ordinary sitz bath, manual flushing sitz bath, electric flushing sitz bath
- electric group (Experimental): Patients in the electric group were advised to use an electric flushing bidet with an irrigator after surgery. The patient was treated with potassium permanganate sitz bath from the first postoperative day. The concentration of potassium permanganate solution used in the sitz bath was 0.02%. The patients were advised to take a sitz bath three times a day (9:00, 13:00, 17:00), and spray potassium permanganate solution in the bidet through an electric douche to achieve the purpose of cleaning the perianal area. The duration of each sitz bath was 10-15 minutes, and the water temperature was 41-43 ° C.
  Interventions: Behavioral: Ordinary sitz bath, manual flushing sitz bath, electric flushing sitz bath

INTERVENTIONS:
Behavioral: Ordinary sitz bath, manual flushing sitz bath, electric flushing sitz bath — Ordinary sitz bath, manual flushing sitz bath, electric flushing sitz bath
  Arms: Manual group; electric group

SUMMARY:
Perianal abscess is a purulent infection of the tissues surrounding the anal canal and rectum. The postoperative wound is prone to infection, and the literature indicates that hip bathing is helpful to prevent infection, reduce edema, and promote healing. Therefore, patients need to use a bidet for medical sitz bath to avoid infection and contamination. The bidet on the market is divided into ordinary type and rinse type (manual or electric). There are no high-quality studies comparing the effects of these sitz baths.

A prospective randomized controlled trial was designed to investigate the effects of regular sitz bath, manual irrigation, and electric irrigation. A total of 102 patients with perianal abscess in the Affiliated Hospital of Putian University were included in the study. The patients were 18-75 years old and underwent surgical treatment. Patients with recurrent abscess, anal fistula, mental disease, pregnant or lactating women, and diabetes were excluded. The patients were divided into general group, manual group and electric group by random number table method, with 34 cases in each group. All patients received hip bathing with 0.02% potassium permanganate solution at 41-43 ° C three times a day for 10-15 minutes each time after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Patients were diagnosed with perianal abscess
* Underwent perianal abscess treatment
* Underwent sitz bath after surgery

Exclusion Criteria:

* Patients with recurrent perianal abscesses or those with concurrent formation of anal fistulas;
* Patients with Crohn's disease;
* Patients with mental disorders;
* Pregnant or lactating women;
* Patients with diabetes;
* Patients with a history of malignant tumor treatment within the past 5 years. ； -Patients who are using immunosuppressants or steroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-08-14 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | Daily from Day 1 until complete epithelialization (max 60 days post-op)
  The effectiveness of different sitbath methods in promoting recovery after perianal abscess was demonstrated by the healing time of the patient's surgical wound.

SECONDARY OUTCOMES:
Complication incidence | Time Frame: Within 30 days postoperatively
  Measurements include the incidence of postoperative bleeding, urinary retention, etc.
pain and swelling | Day 1, 3, 5, 7, and Day 14±2
  visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Putian University Affiliated Hospital, Putian, China

IPD SHARING:
Plan to Share IPD: No